CLINICAL TRIAL: NCT03055806
Title: A Phase 2b, 8-Week, Double-Blind, Placebo-Controlled, Parallel-Group Study to Evaluate the Effects of 3 Different Dose Levels of IX-01 on Intravaginal Ejaculatory Latency Time (IELT), Patient-Reported Outcomes, and Safety in Men With Lifelong Premature Ejaculation (PE)
Brief Title: IX-01 Effect on Intravaginal Ejaculatory Latency Time (IELT), Patient Reported Outcomes and Safety in Men With Premature Ejaculation (PE)
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Ixchelsis Limited (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: IX-0105
Record Dates: First submitted 2017-02-14; First posted 2017-02-16 (Actual); Results first posted 2019-10-07 (Actual); Last update posted 2019-10-07 (Actual); Status verified 2019-03

CONDITIONS: Premature Ejaculation
Keywords: Sex; Sexual Dysfunction; IX-01
MeSH Terms: conditions — Premature Ejaculation; Coitus; Sexual Dysfunction, Physiological

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (4):
- IX-01 1200 mg (Experimental): 1200 mg dose comprising three 400 mg caplets administered orally at least 1 hour before or after food and 1-6 hours prior to sexual activity
  Interventions: Drug: IX-01 1200 mg
- Placebo (Placebo Comparator): Three placebo caplets administered orally at least 1 hour before or after food and 1-6 hours prior to sexual activity
  Interventions: Drug: Placebo
- IX-01 800 mg (Experimental): 800 mg dose comprising two 400 mg caplets and one placebo caplet administered orally at least 1 hour before or after food and 1-6 hours prior to sexual activity
  Interventions: Drug: Placebo; Drug: IX-01 800 mg
- IX-01 400 mg (Experimental): 400 mg dose comprising one 400 mg caplet and two placebo caplets administered orally at least 1 hour before or after food and 1-6 hours prior to sexual activity
  Interventions: Drug: IX-01 400 mg; Drug: Placebo

INTERVENTIONS:
Drug: IX-01 400 mg — IX-01 400 mg caplet
  Arms: IX-01 400 mg
Drug: Placebo — Placebo caplet(s)
  Arms: IX-01 400 mg; IX-01 800 mg; Placebo
Drug: IX-01 800 mg — IX-01 800 mg (Two 400 mg caplets)
  Arms: IX-01 800 mg
Drug: IX-01 1200 mg — IX-01 1200 mg (Three 400 mg caplets)
  Arms: IX-01 1200 mg

SUMMARY:
A Phase 2b, 8-week, double-blind, placebo-controlled, parallel group study to evaluate the effect of 3 different dose levels of IX-01 on IELT and patient-reported outcome in men with lifelong PE.

Men with self-reported lifelong PE (International Society for Sexual Medicine (ISSM) definition) and in stable heterosexual relationship will undergo a 4-week run-in period during which they will be asked to attempt intercourse at least 4 times. Men with IELT ≤ 1 minute on at least 75% of attempts at intercourse during the no-treatment run-in period will be randomized for the double-blind phase of the study.

In the double-blind phase of the study, men will be asked to take study drug 1 to 6 hours prior to sexual activity. Men and partners will be asked to attempt intercourse a minimum of 8 times during the 8 week double-blind study treatment. The patient or partner will record the IELT on each occasion by use of a stopwatch.

ELIGIBILITY:
Inclusion Criteria:

1. Men aged ≥18 years and ≤60 years in stable (≥6 months) heterosexual relationship and who have lifelong PE.
2. Premature ejaculation ≤1 minute on ≥75% attempts at sexual intercourse during the run-in period.
3. Meets other aspects of ISSM definition.
4. Patient and partner willing to attempt intercourse at least 4 times during the run-in period and at least 8 additional times during the double-blind part of the study.
5. Partner not planning pregnancy and willing to use contraception (unless not of childbearing potential, e.g, surgically sterilized).
6. Willing to limit use of alcohol on days in which he takes study drug.
7. Capable of giving written informed consent.

Exclusion Criteria:

1. IELT value >2 minutes during the run-in period.
2. <4 attempts at sexual intercourse during the run-in period.
3. Any patient who rates his control of ejaculation as fair, good, or very good.
4. Any patient who rates his ejaculation-related "personal distress" as "not at all" or "a little bit".
5. Erectile Dysfunction.
6. Concomitant use of phosphodiesterase type 5 (PDE5) inhibitors, selective serotonin reuptake inhibitor (SSRIs)/selective serotonin norepinephrine reuptake inhibitor (SSNRIs), monoamine oxidase inhibitors, alpha blockers, 5-alpha reductase inhibitors, topical anesthetics, and/or tramadol.
7. History (last 6 months) of use of Botox or similar product to treat PE.
8. Has received IX-01 in a previous clinical study.
9. Unwilling to stop other treatments for PE (including but not limited to pharmacological, sex therapy, psychotherapy multiple condoms, and prior masturbation).
10. Any other sexual disorder of patient or partner that could interfere with results.
11. Any current sexually transmitted disease.
12. Any major medical condition of patient that could interfere with ability to have sexual activity and/or require hospital treatment.
13. Body mass index (BMI) >40 kg/m2 or weight <60 kg.
14. Participation in a clinical drug study anytime during the 30 days prior to screening.
15. Human immunodeficiency virus (HIV), hepatitis B.
16. History of prostate disease or clinically significant prostate disease.
17. History of myocardial infarction, coronary bypass surgery, coronary artery angioplasty, unstable angina, clinically evident congestive heart failure, cardiac pacemaker, or cerebrovascular accident.
18. Known or suspected history of significant cardiac arrhythmias.
19. History of drug-induced allergic reactions including skin reactions.
20. Significant psychiatric disease and/or risk of suicidal tendency.
21. History of or other evidence of recent alcohol or drug abuse.

Ages: 18 Years to 60 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult
Gender Based: Yes
Enrollment: 239 (Actual)
Dates: Start 2017-02-28 (Actual); Primary Completion 2017-11-17 (Actual); Study Completion 2017-12-06 (Actual)

CONTACTS AND LOCATIONS:
Locations (29):
- United States (29):
  - Coastal Clinical Research Inc, Mobile, Alabama
  - Radiant Research, Inc. - Phoenix SE, Chandler, Arizona
  - Desert Clinical Research, LLC - Radiant, Mesa, Arizona
  - Family Practice Specialists - Radiant, Phoenix, Arizona
  - San Diego Sexual Medicine, San Diego, California
  - Columbine Family Practice - Radiant, Littleton, Colorado
  - South Florida Medical Research Inc., Aventura, Florida
  - A G A Clinical Trials, Hialeah, Florida
  - Clinical Research Center of Florida, Pompano Beach, Florida
  - Center for Marital and Sexual Health of South Florida, West Palm Beach, Florida
  - Northwest Behavioral Research Center, Roswell, Georgia
  - Boston Clinical Trials Inc, Boston, Massachusetts
  - Mens Health Boston, Chestnut Hill, Massachusetts
  - Center For Pharmaceutical Research, Kansas City, Missouri
  - Clifford J Molin MD LTD - Radiant, Las Vegas, Nevada
  - Accumed Research Associates, Garden City, New York
  - Drug Trials America, Hartsdale, New York
  - Manhattan Medical Research, New York, New York
  - Radiant Research, Inc. - Akron, Akron, Ohio
  - Radiant Research, Inc. - Cincinnati, Cincinnati, Ohio
  - Radiant Research, Inc. - Columbus, Columbus, Ohio
  - Urologic Consultants of Southeastern Pennsylvania, Bala-Cynwyd, Pennsylvania
  - Miriam Hospital / The Men's Health Center, Providence, Rhode Island
  - Radiant Research, Inc. - Anderson, Anderson, South Carolina
  - Radiant Research, Inc. - Greer, Greer, South Carolina
  - Radiant Research, Inc. - Dallas, Dallas, Texas
  - Clinical Trials of Texas Incorporated, San Antonio, Texas
  - Radiant Research Inc - San Antonio, San Antonio, Texas
  - Radiant Research, Inc. - Salt Lake City, Murray, Utah

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Althof S, Osterloh IH, Muirhead GJ, George K, Girard N; PEDRIX Multi-Centre Study Group. The Oxytocin Antagonist Cligosiban Fails to Prolong Intravaginal Ejaculatory Latency in Men with Lifelong Premature Ejaculation: Results of a Randomized, Double-Blind, Placebo-Controlled Phase IIb trial (PEDRIX). J Sex Med. 2019 Aug;16(8):1188-1198. doi: 10.1016/j.jsxm.2019.05.015. PMID 31351660

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Placebo | IX-01 400 mg | IX-01 800 mg | IX-01 1200 mg
Started | 48 | 48 | 71 | 72
Completed | 42 | 41 | 58 | 57
Not Completed | 6 | 7 | 13 | 15
Not completed — Adverse Event | 0 | 0 | 1 | 1
Not completed — Lost to Follow-up | 0 | 3 | 6 | 7
Not completed — Physician Decision | 1 | 0 | 0 | 1
Not completed — Protocol Violation | 1 | 0 | 0 | 0
Not completed — Withdrawal of consent to continue drug | 1 | 1 | 2 | 0
Not completed — Withdrawal of consent to continue study | 2 | 3 | 4 | 6
Not completed — Partner not willing to try intercourse | 1 | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Placebo | IX-01 400 mg | IX-01 800 mg | IX-01 1200 mg | Total
Number analyzed (Participants) | 46 | 48 | 68 | 69 | 231
Age, Continuous [Mean (Standard Deviation); unit: years] | 40.2 (9.13) | 41.8 (9.28) | 40.1 (9.78) | 43.8 (8.63) | 41.6 (9.29)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0 | 0 | 0 | 0 | 0
  Male | 46 | 48 | 68 | 69 | 231
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 7 | 5 | 11 | 19 | 42
  Not Hispanic or Latino | 39 | 43 | 57 | 50 | 189
  Unknown or Not Reported | 0 | 0 | 0 | 0 | 0
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Race: White | 40 | 35 | 58 | 57 | 190
  Race: Black or African American | 4 | 8 | 7 | 8 | 27
  Race: Asian | 1 | 2 | 2 | 2 | 7
  Race: American Indian or Alaska Native | 0 | 0 | 1 | 0 | 1
  Race: Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0 | 0
  Race: Other | 1 | 3 | 0 | 2 | 6
Region of Enrollment [Number; unit: participants]
  United States | 46 | 48 | 68 | 69 | 231

OUTCOME MEASURES:

1. Primary Outcome: Change From Baseline in Geometric Mean (GM) Intravaginal Ejaculatory Latency Time (IELT) Over the Treatment Assessment Period
Description: Intravaginal ejaculatory latency time (IELT) was defined as the time from the initiation of sexual intercourse (penetration) until ejaculation occurred and was recorded by the patient or partner using the stopwatch provided.
Time Frame: Last 4 weeks of treatment compared to baseline
Population: Results presented for modified Intent to treat (mITT) population (all randomized participants who took at least 1 dose of study drug and had at least 2 postbaseline nonmissing IELT assessments).
Measure: Least Squares Mean (Standard Error); unit: Seconds
Arm/Group | Placebo | IX-01 400 mg | IX-01 800 mg | IX-01 1200 mg
Number analyzed (Participants) | 46 | 46 | 65 | 64
Seconds | 42.6 (10.9) | 39.7 (10.6) | 44.5 (9.0) | 29.2 (9.1)

2. Secondary Outcome: Fold Change From Baseline in Geometric Mean (GM) IELT Over the Treatment Assessment Period Compared With Baseline
Description: Intravaginal Ejaculatory Latency Time (IELT) was defined as the time from the initiation of sexual intercourse (penetration) until ejaculation occurred and was recorded using the stopwatch provided.
Time Frame: Last 4 weeks of treatment compared to baseline
Population: as for outcome 1
Measure: Least Squares Mean (Standard Error); unit: Fold change
Arm/Group | Placebo | IX-01 400 mg | IX-01 800 mg | IX-01 1200 mg
Number analyzed (Participants) | 46 | 46 | 65 | 64
Fold change | 1.77 (0.11) | 1.56 (0.11) | 1.79 (0.09) | 1.54 (0.09)

3. Secondary Outcome: Proportion of Patients With ≥2.5-fold Increase in Geometric Mean (GM) Intravaginal Ejaculatory Latency Time (IELT) Over the Treatment Assessment Period Compared With Baseline
Description: Intravaginal Ejaculatory Latency Time (IELT) was defined as the time from the initiation of sexual intercourse (penetration) until ejaculation occurred and was measured using the stopwatch provided.
Time Frame: Last 4 weeks of treatment compared to baseline
Population: as for outcome 1
Measure: Number; unit: Proportion of participants
Arm/Group | Placebo | IX-01 400 mg | IX-01 800 mg | IX-01 1200 mg
Number analyzed (Participants) | 46 | 46 | 65 | 64
Proportion of participants | 0.30 | 0.20 | 0.26 | 0.20

4. Secondary Outcome: Proportion of Patients Rating Their Premature Ejaculation (PE) as Improved Per the Clinical Global Impression of Change (CGIC) Questionnaire
Description: 7 point scale ranging from much worse (-3) to much better (3). The proportion refers to the proportion of patients who had the best 2 possible responses [better (2) or much better (3)] on this scale.
Time Frame: Baseline to the end of treatment (approximately 8 weeks)
Population: as for outcome 1
Measure: Number; unit: Proportion of participants
Arm/Group | Placebo | IX-01 400 mg | IX-01 800 mg | IX-01 1200 mg
Number analyzed (Participants) | 46 | 46 | 65 | 64
Proportion of participants
  Better | 0.12 | 0.05 | 0.07 | 0.07
  Much better | 0 | 0.02 | 0.12 | 0

5. Secondary Outcome: Proportion of Patients Achieving Mean Change in Category of ≥1 or ≥2 on Control of Timing of Ejaculation on the Premature Ejaculation Profile (PEP) Questionnaire.
Description: Reported in electronic diary and based on the Premature Ejaculation Profile (PEP). PEP is scored on a 5 point scale with the scores ranging from 0 (worst answer) to 4 (best answer). A mean change in category of ≥1 or ≥2 corresponds to improving control from 'very poor' to 'fair', 'good', or 'very good'; or from 'poor' to 'fair', 'good', or 'very good'.
Time Frame: Baseline to the end of treatment (approximately 8 weeks)
Population: as for outcome 1
Measure: Number; unit: Proportion of participants
Arm/Group | Placebo | IX-01 400 mg | IX-01 800 mg | IX-01 1200 mg
Number analyzed (Participants) | 43 | 44 | 61 | 62
Proportion of participants | 0.35 | 0.18 | 0.33 | 0.18

6. Secondary Outcome: Proportion of Patients Achieving Mean Change in Category of ≥1 or ≥2 in Ejaculation-related Personal Distress on the Premature Ejaculation Profile (PEP) Questionnaire
Description: Reported in e-diary. Based on Premature Ejaculation Profile (PEP). Scale ranges from 'extremely' (0) to 'not at all' (4). An increase in score from baseline indicates improvement. A change in category of ≥1 or ≥2 corresponds to improving distress from 'extremely' to 'moderately', 'a little bit' or 'not at all'; or from 'quite a bit' to 'moderately', 'a little bit' or 'not at all'; or from 'moderately' to 'a little bit' or 'not at all'.
Time Frame: Baseline to the end of treatment (approximately 8 weeks)
Population: as for outcome 1
Measure: Number; unit: Proportion of participants
Arm/Group | Placebo | IX-01 400 mg | IX-01 800 mg | IX-01 1200 mg
Number analyzed (Participants) | 43 | 44 | 61 | 62
Proportion of participants | 0.37 | 0.25 | 0.39 | 0.23

7. Secondary Outcome: Proportion of Patients Achieving Change in Category of ≥2 on Control of Timing of Ejaculation and Achieving Change in Category of ≥1 in Ejaculation-related Personal Distress at End of Treatment
Description: Reported in electronic diary and based on the Premature Ejaculation Profile (PEP). PEP is scored on a 5 point scale with the scores ranging from 0 (worst answer) to 4 (best answer).
Time Frame: Baseline to the end of treatment (approximately 8 weeks)
Population: as for outcome 1
Measure: Number; unit: Proportion of participants
Arm/Group | Placebo | IX-01 400 mg | IX-01 800 mg | IX-01 1200 mg
Number analyzed (Participants) | 46 | 46 | 65 | 64
Proportion of participants | 0.13 | 0.11 | 0.25 | 0.08

8. Secondary Outcome: Mean Change From Baseline in Score on Control of Ejaculation
Description: Reported in electronic diary and based on the Premature Ejaculation Profile (PEP). PEP question on control of timing is scored on a 5 point scale with the scores ranging from very poor (this is the worst answer scored as 0) to very good (this is the best answer scored as 4).
Time Frame: Last 4 weeks of treatment compared to baseline
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Placebo | IX-01 400 mg | IX-01 800 mg | IX-01 1200 mg
Number analyzed (Participants) | 46 | 46 | 65 | 64
score on a scale | 0.55 (0.938) | 0.46 (0.837) | 0.58 (0.868) | 0.32 (0.619)

9. Secondary Outcome: Mean Change From Baseline in Score on Ejaculation-related Personal Distress
Description: Based on Premature Ejaculation Profile (PEP). Scale ranges from 'extremely' (0) to 'not at all' (4). An increase in score from baseline indicates improvement.
Time Frame: Last 4 weeks of treatment compared to baseline
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Placebo | IX-01 400 mg | IX-01 800 mg | IX-01 1200 mg
Number analyzed (Participants) | 46 | 46 | 65 | 64
score on a scale | 0.73 (1.139) | 0.38 (1.036) | 0.58 (0.933) | 0.51 (0.898)

ADVERSE EVENTS:
Time Frame: Adverse event data were collected from Baseline (Week 0) to the Follow-Up visit (Week 10).
Arm/Group | Placebo | IX-01 400 mg | IX-01 800 mg | IX-01 1200 mg
All-Cause Mortality (participants affected / at risk) | 0/46 | 0/48 | 0/68 | 0/69
Serious Adverse Events (participants affected / at risk) | 0/46 | 0/48 | 0/68 | 0/69
Other Adverse Events (participants affected / at risk) | 12/46 | 8/48 | 12/68 | 18/69
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Placebo (N=46) | IX-01 400 mg (N=48) | IX-01 800 mg (N=68) | IX-01 1200 mg (N=69)
Dizziness (Nervous system disorders) | 0 | 0 | 0 | 1
Headache (Nervous system disorders) | 3 | 2 | 2 | 2
Hypersomnia (Nervous system disorders) | 0 | 0 | 1 | 0
Memory impairment (Nervous system disorders) | 0 | 0 | 0 | 1
Parosmia (Nervous system disorders) | 1 | 0 | 0 | 0
Poor quality sleep (Nervous system disorders) | 0 | 1 | 0 | 0
Bronchitis (Infections and infestations) | 0 | 0 | 0 | 1
Gastroenteritis (Infections and infestations) | 0 | 0 | 1 | 0
Nasopharyngitis (Infections and infestations) | 1 | 1 | 1 | 2
Otitis media (Infections and infestations) | 0 | 1 | 0 | 0
Tinea cruris (Infections and infestations) | 0 | 0 | 0 | 1
Upper respiratory tract infection (Infections and infestations) | 2 | 0 | 1 | 0
Abnormal dreams (Psychiatric disorders) | 1 | 0 | 0 | 1
Depressed mood (Psychiatric disorders) | 1 | 0 | 0 | 0
Insomnia (Psychiatric disorders) | 0 | 1 | 1 | 0
Libido decreased (Psychiatric disorders) | 0 | 1 | 1 | 0
Libido increased (Psychiatric disorders) | 0 | 1 | 0 | 0
Blood potassium increased (Investigations) | 0 | 0 | 1 | 0
Blood pressure increased (Investigations) | 1 | 0 | 0 | 0
Haematocrit increased (Investigations) | 0 | 0 | 0 | 1
Neutrophil count increased (Investigations) | 0 | 0 | 0 | 1
Red blood cell count increased (Investigations) | 0 | 0 | 0 | 1
Red blood cells urine positive (Investigations) | 0 | 1 | 0 | 0
Weight decreased (Investigations) | 0 | 0 | 1 | 0
White blood cell count increased (Investigations) | 0 | 0 | 0 | 1
Abdominal pain (Gastrointestinal disorders) | 0 | 0 | 1 | 0
Abdominal pain upper (Gastrointestinal disorders) | 0 | 0 | 0 | 1
Dry mouth (Gastrointestinal disorders) | 0 | 0 | 0 | 1
Dyspepsia (Gastrointestinal disorders) | 0 | 1 | 0 | 0
Faeces discoloured (Gastrointestinal disorders) | 0 | 0 | 0 | 1
Concussion (Injury, poisoning and procedural complications) | 1 | 0 | 0 | 0
Laceration (Injury, poisoning and procedural complications) | 0 | 0 | 1 | 1
Ligament sprain (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 1
Skin abrasion (Injury, poisoning and procedural complications) | 1 | 0 | 0 | 0
Stress fracture (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 1
Arthralgia (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1 | 0
Back pain (Musculoskeletal and connective tissue disorders) | 1 | 0 | 1 | 0
Joint hyperextension (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 1
Myalgia (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0 | 0
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1 | 0
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 2
Rhinitis allergic (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 1
Asthenia (General disorders) | 0 | 0 | 0 | 1
Energy increased (General disorders) | 0 | 0 | 0 | 1
Fatigue (General disorders) | 0 | 1 | 0 | 0
Pyrexia (General disorders) | 0 | 1 | 0 | 0
Erectile dysfunction (Reproductive system and breast disorders) | 1 | 0 | 1 | 1
Diabetes mellitus (Metabolism and nutrition disorders) | 1 | 0 | 0 | 0
Hyperkalaemia (Metabolism and nutrition disorders) | 0 | 0 | 1 | 0
Hypertension (Vascular disorders) | 0 | 0 | 1 | 1
Angina pectoris (Cardiac disorders) | 0 | 0 | 1 | 0
Cholelithiasis (Hepatobiliary disorders) | 0 | 0 | 1 | 0
Rash maculo-papular (Skin and subcutaneous tissue disorders) | 0 | 0 | 1 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Sponsor may chose to collaborate on authorship, and sponsor's agent has 60-day review.

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2017-01-16): https://cdn.clinicaltrials.gov/large-docs/06/NCT03055806/Prot_SAP_000.pdf